CLINICAL TRIAL: NCT05963854
Title: An Innovative, Accessible, and Flexible Approach for Household Food Waste Measurement
Brief Title: Food Survey, Curbside, Remote APPs SC
Acronym: Food SCRAPPsSC
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Martin, Corby, K., M.D. (Individual)
Responsible Party: Principal Investigator, John Apolzan, Associate Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-007 A
Record Dates: First submitted 2023-07-14; First posted 2023-07-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Waste Management; Recycling; Climate; Nutrition Sciences

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SC: Food Waste Tracking Survey and Curbside over 2 consecutive weeks
  Interventions: Other: Survey Curbside

INTERVENTIONS:
Other: Survey Curbside — Observational. Waste will be collected on specific days for 2 consecutive weeks and surveys will be completed to coincide with the waste collections.
  Other Names: SC

SUMMARY:
The proposed research will create accurate and standardized household FW measurement methodologies that foster serial and longitudinal assessments as well as confident and convenient one-time measurement by stakeholders. The investigators will have participants simutaneously deploy (1) retrospective surveys (2) curbside audits.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, age 18 years and older
* Willing and able to store household food waste for curbside pickup by a third-party waste pickup company
* Internet or Wi-Fi availability to complete online surveys

Exclusion Criteria:

* Not willing to adhere to study procedures and study visit timelines
* Any condition or circumstance that in the judgement of the PI could interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the greater Columbus, OH and Baton Rouge, LA regions.
Sampling Method: Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Total Household Food Waste | 1 week
  Weight

SECONDARY OUTCOMES:
Household Food Waste Energy | 1 week
  Energy (kcal)

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication after a DTA with the institution. Please provide research question to investigators.
Supporting Information: Study Protocol, ICF